CLINICAL TRIAL: NCT00252863
Title: A Comparison of Symbicort Single Inhaler Therapy (Symbicort Turbuhaler 160/4.5 µg, 1 Inhalation b.i.d. Plus as Needed) and Conventional Best Practice for the Treatment of Persistent Asthma in Adults - a 26-Week, Randomised, Open-Label, Parallel-Group, Multicentre Study
Brief Title: DESOLO - SiT Peri-Launch: A Comparison of Symbicort Single Inhaler Therapy and Conventional Best Practice for the Treatment of Persistent Asthma in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5890L00011; DESOLO
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Health Services Needs and Demand; Budesonide; Fluticasone; Theophylline; montelukast

INTERVENTIONS:
Drug: Symbicort, used twice daily (b.i.d) and as needed (prn)
Drug: Budesonide Turbuhaler 200 µg
Drug: Fluticasone Discus 250 µg
Drug: Formoterol Turbuhaler 4.5 µg
Drug: Terbutaline Turbuhaler 0.5 mg
Drug: Salbutamol pressurized metered dose inhaler (pMDI) 100 µg
Drug: Salmeterol Discus 50 µg
Drug: Budesonide/Formoterol Turbuhaler 160/4.5 µg
Drug: Fluticasone/Salmeterol Discus 250/50 µg
Drug: Fluticasone/Salmeterol Discus 500/50 µg
Drug: Theophylline 200 mg
Drug: Theophylline 300 mg
Drug: Singulair 10 mg

SUMMARY:
The purpose of this study is to determine whether Symbicort dosed according to the Symbicort Maintenance and Reliever Therapy (SMART) concept is superior to standard asthma treatment according to the local German treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with asthma, either well-controlled on a regular therapy with a combination of long-acting beta-agonists and inhaled corticosteroids or symptomatic on therapy with inhaled corticosteroids alone.

Exclusion Criteria:

* Any other significant lung disease other than asthma
* Any disease that might put patients at risk if they participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600
Dates: Start 2004-12; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Time to first severe asthma exacerbation

SECONDARY OUTCOMES:
Number of severe asthma exacerbations
Mean use of as-needed medication
Change in forced expiratory volume in 1 second (FEV1) from the end of run-in to the end of the study period
Prescribed asthma medication during the treatment period
Asthma Control Questionnaire (ACQ)
Patient's satisfaction with the treatment question
Health care contacts
Asthma medication
Time lost from paid and unpaid work
Serious adverse events (SAEs)
Discontinuations due to adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Worth, MD, Principal Investigator — Klinikum Fürth
Locations (169):
- Germany (169):
  - Research Site, Stuttgart, Baden-Wurttemberg
  - Research Site, München, Bavaria
  - Research Site, Cottbus, Brandenburg
  - Research Site, Hamburg, Hamburg
  - Research Site, Frankfurt am Main, Hesse
  - Research Site, Hanover, Lower Saxony
  - Research Site, Rostock, Mecklenburg-Vorpommern
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Münster, North Rhine-Westphalia
  - Research Site, Mainz, Rhineland-Palatinate
  - Research Site, Saarbrücken, Saarland
  - Research Site, Dresden, Saxony
  - Research Site, Halle, Saxony-Anhalt
  - Research Site, Bad Segeberg, Schleswig-Holstein
  - Research Site, Berlin, State of Berlin
  - Research Site, Jena-Maua, Thuringia
  - Research Site, Amberg
  - Research Site, Aschaffenburg
  - Research Site, Auerbach
  - Research Site, Augsburg
  - Research Site, Backnang
  - Research Site, Bad Arolsen
  - Research Site, Bad Doberan
  - Research Site, Bad Lippspringe
  - Research Site, Bad Neuenahr
  - Research Site, Bad Reichenhall
  - Research Site, Bad Sessendorf
  - Research Site, Bayreuth
  - Research Site, Bensheim
  - Research Site, Bergisch Gladbach
  - Research Site, Berlin
  - Research Site, Bitte Eintragen
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Borna
  - Research Site, Brake
  - Research Site, Burg
  - Research Site, Burgwedel
  - Research Site, Castrop-Rauxel
  - Research Site, Chemnitz
  - Research Site, Cologne
  - Research Site, Coswig
  - Research Site, Cottbus
  - Research Site, Damme
  - Research Site, Darmstadt
  - Research Site, Deggendorf
  - Research Site, Dillingen
  - Research Site, Dinslaken
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Dülmen
  - Research Site, Düsseldorf
  - Research Site, Eisenach
  - Research Site, Eisenhüttenstadt
  - Research Site, Emden
  - Research Site, Erfurt
  - Research Site, Erkelenz
  - Research Site, Eschwege
  - Research Site, Flensburg
  - Research Site, Forchheim
  - Research Site, Frankenthal
  - Research Site, Frankfurt
  - Research Site, Freiberg
  - Research Site, Freiburg im Breisgau
  - Research Site, Freising
  - Research Site, Fulda
  - Research Site, Fürstenwalde
  - Research Site, Fürth
  - Research Site, Gelsenkirchen
  - Research Site, Giessen
  - Research Site, Gotha
  - Research Site, Göppingen
  - Research Site, Günzburg
  - Research Site, Gütersloh
  - Research Site, Hagen
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hamm
  - Research Site, Hanover
  - Research Site, Harpstedt
  - Research Site, Hartha
  - Research Site, Heidelberg
  - Research Site, Heilbronn
  - Research Site, Homburg-Saar
  - Research Site, Hoyerswerda
  - Research Site, Iserloh
  - Research Site, Kamen
  - Research Site, Kamenz
  - Research Site, Kamp-Lintfort
  - Research Site, Karlsruhe
  - Research Site, Kassel
  - Research Site, Kaufbeuren
  - Research Site, Kempten
  - Research Site, Kiel
  - Research Site, Kitzingen
  - Research Site, Koblenz
  - Research Site, Krefeld
  - Research Site, Kronach
  - Research Site, Landsberg
  - Research Site, Leipzig
  - Research Site, Leonberg
  - Research Site, Leverkusen
  - Research Site, Loerrach
  - Research Site, Ludwigsburg
  - Research Site, Lübeck
  - Research Site, Lüneburg
  - Research Site, Magdeburg
  - Research Site, Mainaschaff
  - Research Site, Mainz
  - Research Site, Marburg
  - Research Site, Markkleeberg
  - Research Site, Memmingen
  - Research Site, Moers
  - Research Site, Mönchengladbach
  - Research Site, Mühlhausen
  - Research Site, München
  - Research Site, Neubrandenburg
  - Research Site, Neuss
  - Research Site, Neuwied
  - Research Site, Niesky
  - Research Site, Nordhausen
  - Research Site, Oberhausen
  - Research Site, Oranienburg
  - Research Site, Oschersleben
  - Research Site, Paderborn
  - Research Site, Passau
  - Research Site, Peine
  - Research Site, Pforzheim
  - Research Site, Pinneberg
  - Research Site, Potsdam
  - Research Site, Ratingen
  - Research Site, Recklinghausen
  - Research Site, Regensburg
  - Research Site, Reutlingen
  - Research Site, Rheine
  - Research Site, Rodenbach
  - Research Site, Rostock
  - Research Site, Rottweil
  - Research Site, Rudolstadt
  - Research Site, Saalfeld
  - Research Site, Saarbrücken
  - Research Site, Saarlouis
  - Research Site, Salzgitter
  - Research Site, Sangerhausen
  - Research Site, Schleswig
  - Research Site, Schwabach
  - Research Site, Schwäbisch Gmünd
  - Research Site, Schwerin
  - Research Site, Siegen
  - Research Site, Simmern
  - Research Site, Sindelfingen
  - Research Site, Singen
  - Research Site, Solingen
  - Research Site, Stade
  - Research Site, Stadthagen
  - Research Site, Steinhagen
  - Research Site, Stuttgart
  - Research Site, Trier
  - Research Site, Ulm
  - Research Site, Uttenreuth
  - Research Site, Wardenburg
  - Research Site, Wedel
  - Research Site, Weinheim
  - Research Site, Weyhe
  - Research Site, Witten
  - Research Site, Worpswede
  - Research Site, Würzburg
  - Research Site, Zerbst
  - Research Site, Zwickau